CLINICAL TRIAL: NCT03530722
Title: Ex-vivo Performance Evaluation of the Histolog™ Scanner for Human Breast Carcinoma Detection on Fresh Breast Core Biopsies
Status: Completed | Type: Observational
Sponsor: Brust-Zentrum AG (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-00836
Record Dates: First submitted 2018-04-19; First posted 2018-05-21 (Actual); Last update posted 2018-05-21 (Actual); Status verified 2018-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Fresh breast core biopsies suspicious for breast cancer that are usually taken during clinical breast assessments will be imaged via confocal microscopy.

The device so called HistologTM Scanner is based on confocal fluorescence and displays microscopic histology images superficial layers of fresh tissue.

After the imaging procedure the fresh breast tissue specimen will be followed according to the gold standard workflow (H&E-stained images).

Subsequently, two pathologists will analyze the HistologTM Scanner obtained-images and H&E-stained images for potential breast cancer structures.

A comparison of both analyses for cancer visualization will be performed to evaluate the feasibility of using confocal microscopy for breast cancer detection.

DETAILED DESCRIPTION:
During clinical breast assessments physicians may detect diagnostic findings suspicious for breast cancer. In such situations a biopsy has to be taken to confirm the diagnosis histologically. Once informed consent will be obtained, the physician will collect a biopsy sample using the standard procedure with US- or MG-guided Biospy. Immediately prior to gold standard pathology workflow (formalin fixation), HistologTM Scanner will be used to image the fresh biopsy specimens. The HistologTM Scanner (v1.0, SamanTree Medical SA, Lausanne, Switzerland, CE marking) is based on confocal fluorescence and displays microscopic histology images of superficial layers of fresh tissue after nuclear staining with Acridine Orange (30 seconds) and rinsing in saline solution.

Finally, the specimen will be processed following the gold standard workflow (H&E-stained images).

Two independent pathologists will assess the HistologTM Scanner- and H&E-stained images subsequently according to the B-classification (categories B1-B5; "0" was defined as "no diagnosis possible") and determine the correspondence of the results.

ELIGIBILITY:
Inclusion Criteria:

* Adult female patient ≥18 years old.
* Patient presenting with suspected breast carcinoma.
* Patient eligible for biopsy sampling.
* Patient must sign a written informed consent prior to research project entry.

Exclusion Criteria:

* Patient previously treated for breast carcinoma.
* Patient has undergone previous neo-adjuvant treatment.
* Patient is not willing to participate in the research project.
* Patient is not capable of consenting.
* Patient is younger than 18 years old
* Patient is male

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult female patients presenting lesions suspicious for breast carcinoma in ultrasound or mammography that are eligible for biopsy sampling and meet the research project's inclusion/exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2017-07-04 (Actual); Primary Completion 2017-11-15 (Actual); Study Completion 2017-12-11 (Actual)

PRIMARY OUTCOMES:
Correspondence of pathologic assessment in specimen suspicious for breast cancer | up to 24 weeks
  Evaluate the correspondence of breast cancer diagnosis based on confocal HistologTM Scanner images in comparison with gold standard pathology assessment.

SECONDARY OUTCOMES:
Usability of the HistologTM Scanner confocal device | up to 24 weeks
  Assess the usability of the HistologTM Scanner confocal device in the context of breast surgery by gathering feedback and expert opinion from the medical staff involved in the research study.
Acceptance of the HistologTM Scanner confocal device | up to 24 weeks
  Assess the acceptance of the HistologTM Scanner confocal device in the context of breast surgery by gathering feedback and expert opinion from the medical staff involved in the research study.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Tausch, MD, Principal Investigator — Brust-Zentrum AG Zürich
Locations (1):
- Brust-Zentrum AG, Zurich, Switzerland